CLINICAL TRIAL: NCT00913900
Title: Stem Cell Revascularization in Patients With Critical Limb Ischemia
Brief Title: Safety Study of Adult Stem Cells to Treat Patients With Severe Leg Artery Disease
Acronym: SCRIPT-CLI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failure to mobilize adequate CD34+ stem cells for minimum study treatment dose.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2009-0008
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Critical Limb Ischemia; Arterial Occlusive Disease; Vascular Diseases
Keywords: Arterial Occlusive Diseases; Vascular Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Stem cells (CD133+) (Active Comparator): Intramuscular injection
  Interventions: Biological: autologous CD133+ cells
- Control (Placebo Comparator): Intramuscular Injection
  Interventions: Biological: autologous CD133+ cells

INTERVENTIONS:
Biological: autologous CD133+ cells — Intramuscular injection

SUMMARY:
Peripheral artery disease (PAD) due to leg artery blockages can result in painful leg muscles, skin ulcers and infection due to poor blood flow. In severe forms, the only treatment may be amputation. Adult stem cells injected into affected legs may cause new blood vessel formation and improve blood flow. The purpose of this study is to determine the feasibility and safety of injecting adult stem cells into the leg muscles of patients with severe PAD, in an attempt to improve blood flow.

DETAILED DESCRIPTION:
Lower extremity peripheral artery disease (PAD) is a common, debilitating and potentially life-threatening illness. Obstructive PAD can progress to limb-threatening ischemia with rest pain, ulcers, and gangrene requiring amputation unless blood flow to the ischemic limb can be restored. Surgical revascularization options are often limited by arteries that are too small to bypass. Patient co-morbidities also make surgical options risky. Percutaneous revascularization techniques are similarly limited by small distal artery caliber, technical difficulty and high restenosis rates. Amputation may be the only treatment option for non-healing ulcers or gangrene. Direct intramuscular injection of adult stem cells may result in improved lower extremity perfusion, symptomatic improvement and limb salvage in patients with critical limb ischemia not optimal for conventional revascularization. This study aims to demonstrate the safety and feasibility of this therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory critical limb ischemia (Rutherford Score 4/5)
* Not optimal for surgical or catheter-based revascularization
* Obstructive atherosclerosis of at least 1 major artery in both limbs
* Ankle-Brachial Index <0.6 or Absolute Ankle pressure <60mmHg or toe pressure <40mmHg or pulse volume recording that is flat or barely pulsatile

Exclusion Criteria:

* Gangrene(Rutherford 6) or pre-existing major tissue loss
* Unstable Angina, MI, stroke, CHF (class III or IV) within 6 months of study treatment

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Death or amputation | 6 months

SECONDARY OUTCOMES:
Vascular hemodynamics and function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amish N Raval, MD, Principal Investigator — U.Wisconsin School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Raval AN, Schmuck EG, Tefera G, Leitzke C, Ark CV, Hei D, Centanni JM, de Silva R, Koch J, Chappell RG, Hematti P. Bilateral administration of autologous CD133+ cells in ambulatory patients with refractory critical limb ischemia: lessons learned from a pilot randomized, double-blind, placebo-controlled trial. Cytotherapy. 2014 Dec;16(12):1720-32. doi: 10.1016/j.jcyt.2014.07.011. Epub 2014 Sep 18. PMID 25239491
- [Derived] Moazzami B, Mohammadpour Z, Zabala ZE, Farokhi E, Roohi A, Dolmatova E, Moazzami K. Local intramuscular transplantation of autologous bone marrow mononuclear cells for critical lower limb ischaemia. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD008347. doi: 10.1002/14651858.CD008347.pub4. PMID 35802393